CLINICAL TRIAL: NCT00841230
Title: Additional Value of Deanxit in Tinnitus Patients Treated With Rivotril
Brief Title: Deanxit and Rivotril in Tinnitus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof Dr P H Van de Heyning, Antwerp University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8/46/260
Record Dates: First submitted 2009-01-30; First posted 2009-02-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — flupentixol, melitracen drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactose placebo (Placebo Comparator): 1x/day
  Interventions: Drug: Lactose placebo
- Deanxit (Experimental)
  Interventions: Drug: Deanxit

INTERVENTIONS:
Drug: Deanxit — Deanxit 1x/day
  Arms: Deanxit
Drug: Lactose placebo — Lactose used as placebo
  Arms: Lactose placebo

SUMMARY:
The purpose of this study is to investigate whether increased tinnitus reduction can be obtained with Deanxit in patients already receiving Rivotril.

ELIGIBILITY:
Inclusion Criteria:

* pure tone, narrow band noise or polyphonic tinnitus
* unilateral or bilateral tinnitus
* VAS ≥ 4

  * cochleair origin tinnitus
  * tinnitus present 3 months or more
  * age 18y or more
  * intake Rivotril 1mg/d
  * patient 'able to cooperate'
  * patient able to fill in TQ en VAS
  * No pontine angle pathology on MRI

Exclusion Criteria:

* pulsatile tinnitus
* pregnancy or breast feeding
* contra-indications Deanxit
* recovery myocard infarct
* conduction disorder His
* untreated glaucoma
* MAO inhibitors: 15d stop
* otosclerosis
* middle ear pathologies
* Ménière
* somatic tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Meeus, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Antwerp, Antwerp, Belgium